CLINICAL TRIAL: NCT00918125
Title: The Use of Educational Videos to Improve Patient Decision Making and Racial Disparities in the Implantation of Implantable Cardioverter Defibrillators (ICDs)
Brief Title: Educational Videos to Improve Patient Decision Making and Race Disparities in Implantable Cardioverter Defibrillator Use
Acronym: VIVID-01
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00011117; 1U18HS016964 (AHRQ)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Results first posted 2013-04-05 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2013-04

CONDITIONS: Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- White educational video: Patients will view an educational video that contains White physicians and patients.
- African-American educational video: Patients will view an educational video that contains African-American physicians and patients.
- Usual care: Patients will receive counseling about their condition and treatment options.

SUMMARY:
The investigators will examine whether an educational video increases patient knowledge about heart failure and the risk of sudden cardiac arrest and leads to greater satisfaction with information provided as compared to usual care. Additionally, the investigators will look at whether racial concordance (physician and patient being of the same race) improves satisfaction with the patient's treatment decision and disease knowledge. Our hypothesis is that a video in which participants are of the same race as the patient will provide better education and more satisfaction with the treatment decision and may lead to more patients choosing ICD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Class I primary prevention indications for an implantable cardioverter defibrillator (ICD). These include:
* Patients with ejection fraction <35% due to prior myocardial infarction (MI) who are at least 40 days post-MI and with New York Heart Association (NYHA) functional class II or III;OR
* Patients with nonischemic dilated cardiomyopathy (DCM) who have an LVEF < 35% and who meet criteria for NYHA functional class II or III; OR
* Patients with left ventricular dysfunction due to prior MI who are at least 40 days post-MI, have an left ventricular ejection fraction (LVEF) <30% and are in NYHA functional class I-III; OR
* Patients with nonsustained ventricular tachycardia (VT) due to prior MI, LVEF <40%, and with inducible ventricular fibrillation (VF) or sustained VT at electrophysiological study; AND
* Self identified race as black/African American or white/Caucasian

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for an implantable cardioverter defibrillator (ICD) for the primary prevention of sudden cardiac death.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Peterson, MD, MPH, Principal Investigator — DCRI
Locations (2):
- United States (2):
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Thomas KL, Zimmer LO, Dai D, Al-Khatib SM, Allen LaPointe NM, Peterson ED. Educational videos to reduce racial disparities in ICD therapy via innovative designs (VIVID): a randomized clinical trial. Am Heart J. 2013 Jul;166(1):157-63. doi: 10.1016/j.ahj.2013.03.031. Epub 2013 May 15. PMID 23816035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 3 centers: Duke University Medical Center, Alamance Regional Hospital; and Southeast Regional Medical Center in North Carolina. Patients were enrolled during 2011.
Groups:
- Standard of Care: Patients in this arm received standard of care (counseling from a physician).
- Video Intervention: Patients in this arm viewed an educational video on sudden cardiac arrest and ICDs.
Period: Overall Study
Arm/Group | Standard of Care | Video Intervention
Started | 20 | 39
Completed | 20 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Black Patients: Patients who self-identified as African American
- White Patients: Patients who self-identified as White
- Total: Total of all reporting groups
Arm/Group | Black Patients | White Patients | Total
Number analyzed (Participants) | 22 | 37 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (11.4) | 61.7 (17.5) | 58.2 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 14 | 23 | 37
Randomization Allocation [Number; unit: participants] — Patients were randomized into three study arms, stratified by race: white video, black video or usual care
  participants
    Video | 15 | 24 | 39
    Usual Care | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Decision to Receive an ICD
Description: At one week post-intervention, patients were asked what treatment option they preferred: ICD placement with medications; No ICD, continue with medications only; or unsure.
Time Frame: 1 week post intervention
Population: All patients with available data at one week
Measure: Number; unit: Participants
Groups:
- Video: All patients who saw an educational video
- Standard of Care: Usual care
Arm/Group | Video | Standard of Care
Number analyzed (Participants) | 39 | 17
Participants | 28 | 14

2. Secondary Outcome: Decisional Conflict Scale
Description: At one week post-intervention, patients were asked 9 questions from a modified decisional conflict scale to assess overall decisional conflict and three subscales (decision uncertainty; factors contributing to uncertainty; and perceived effective decision making). Overall scores range from 9 (no decisional conflict) to 45 (high decisional conflict).
Time Frame: one week post intervention
Population: Patients with data at one week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video | Standard of Care
Number analyzed (Participants) | 39 | 14
units on a scale | 35.0 (2.9) | 34.1 (3.5)

3. Secondary Outcome: Receipt of an ICD
Description: Patients were asked (or medical records reviewed) to determine if patients did receive an ICD within approximately 3 months post intervention.
Time Frame: 3 months
Population: All patients with data at 3 months
Measure: Number; unit: participants
Groups:
- African Americans: African Americans in study from all study arms
- Whites: Whites in study from all study arms
Arm/Group | African Americans | Whites
Number analyzed (Participants) | 22 | 37
participants | 14 | 33

4. Other Pre Specified Outcome: Mean Knowledge Scores About ICD Therapy One Week Post Intervention.
Description: We assessed knowledge of ICD therapy prior to the educational intervention, directly after the educational intervention and one week later. The tool used was a 13 question tool on key aspects of ICDs, risks and benefits, and health conditions eligible for an ICD. Scores could range from 0-13, with higher score indicating greater levels of knowledge.
Time Frame: one week post intervention
Population: Mean scores were calculated with one point for each correct answer out of 13 questions for all patients with data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- African Americans: All African Americans in study
- Whites: All Whites in study
Arm/Group | African Americans | Whites
Number analyzed (Participants) | 22 | 37
units on a scale | 9.9 (2.5) | 10.4 (3.0)

ADVERSE EVENTS:
Time Frame: No adverse events were collected for this study, which was a purely educational intervention.
Groups:
- All Patients: Patients in this arm received standard of care (counseling from a physician).
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study terminated early and thus only 59 out of the proposed 90 patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No